CLINICAL TRIAL: NCT04941443
Title: Methadone for Pain Relief in First Trimester Medication Abortion
Brief Title: Methadone and Medication Abortion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit more participants.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-41109
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-12

CONDITIONS: Pain; Medical Abortion
Keywords: Oral methadone; Pain control
MeSH Terms: conditions — Pain; Agnosia | interventions — Methadone; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oral methadone (Experimental): Participants will be given a preemptive analgesic in addition to a standard dose of ibuprofen while undergoing early medication abortion with mifepristone and misoprostol (not provided as part of the study). All participants will also be provided with supplementary non- opioid analgesics to be used at their own discretion during the process.
  Interventions: Drug: Methadone Pill; Drug: Ibuprofen

INTERVENTIONS:
Drug: Methadone Pill — All participants will be given a 5mg methadone tablet to be taken immediately following the misoprostol dose.
  Other Names: Methadone Hydrochloride
Drug: Ibuprofen — All participants will be provided additional analgesics (ibuprofen 800mg x4 tabs) available for use as needed every eight hours.
  Other Names: Motrin, Advil

SUMMARY:
Pain has been recognized to be the most common and predictable side effect of medication abortion, causing significant distress associated with the process. Yet there is little known about the appropriate management of pain during this process, with no current evidence based recommendations for optimal analgesic regimens during the first trimester.

The goal of this study is to evaluate the efficacy of oral methadone for pain control during medication abortion. The current medication regimen used to perform medication abortion is a dose of mifepristone (antiprogesterone) orally, followed by a dose of misoprostol (prostaglandin analogue) 24 to 72 hours later. Patients are prescribed a standard dose of ibuprofen 600-800mg tabs for pain control during the process. The investigators will conduct a non-randomized, pilot study with 25 patients evaluated at the Boston Medical Center family planning clinic at 10 weeks of gestation or less for medication abortion.

DETAILED DESCRIPTION:
The primary objective of this research study is to determine the feasibility of enrolling patients in a study that requires the consumption of methadone for acute pain management for medication abortion. Secondary objectives include the assessment of pain using: pain scores at 0, 4, 8, and 24 hours following misoprostol, use of supplementary analgesia, reported side effects, and patient satisfaction

All participants will be instructed to take methadone 5 mg orally (1 tablet) simultaneously with the consumption of misoprostol. The participants will be evaluated using an 11 point numeric rating pain scale with 0 (no pain) and 10 (most severe pain). Patients will be given a telephone number to which they will be asked to text study staff indicating that misoprostol and methadone have been consumed. Study staff will phone the participants at 0, 4, 8 and 24 hours post misoprostol consumption to conduct a survey posing questions about maximum pain scores, compliance with study medication and any adverse effects experienced. Participants will also be contacted at 48 hours for further evaluation of any reported adverse events and 1 week post misoprostol to assess ease of study design and instructions, pain experience, perisomal view on consumption of methadone and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women requesting medication abortion up to 10 weeks gestation
* Fluent English speaking
* Able and willing to receive and send text messages and receive phone calls
* Opioid naive
* Healthy patients with no significant comorbidities

Exclusion Criteria:

* Any history of drug or alcohol use, opioid use in last 30 days, chronic use of pain medications, or use of benzodiazepines.
* Any chronic disease including renal, liver, respiratory or cardiac disease
* Any known allergies to mifepristone, misoprostol, nonsteroidal anti-inflammatory drugs (such as ibuprofen) and methadone.
* Known history of QT prolongation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Achu, MD, Principal Investigator — Boston Medical Center, Anesthesiology Department
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Methadone
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Oral Methadone
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 24 Hours Post Medication Abortion
Description: Pain will be assessed using measured by an 11-point numeric visual analogue (VAS); (0-10) where 0 is equivalent to no pain and 10 is the worst pain. Higher scores are associated with more pain.
Time Frame: 24 hours
Population: Of the 4 consented participants, none provided the information needed for any of the outcome measures, so no results are available.
Arm/Group | Oral Methadone
Number analyzed (Participants) | 0

2. Secondary Outcome: Pain Score at 8 Hours Post Medication Abortion
Description: as for outcome 1
Time Frame: 8 hours
Population: as for outcome 1
Arm/Group | Oral Methadone
Number analyzed (Participants) | 0

3. Secondary Outcome: Participant Satisfaction
Description: An investigator developed survey will be administered over the phone by study staff to assess participant satisfaction. Participants will be asked how satisfied they were with their pain management and a Likert scale will be used to collect responses. The response choices range from 0= very dissatisfied to 4= very satisfied.
Time Frame: 24 hours, 1 week
Population: as for outcome 1
Arm/Group | Oral Methadone
Number analyzed (Participants) | 0

4. Secondary Outcome: Adverse Events
Description: An investigator developed survey will be administered over the phone by study staff to assess adverse events including dizziness, difficulty breathing, nausea or vomiting.
Time Frame: 24 hours, 48 hours, 1 week
Population: as for outcome 1
Arm/Group | Oral Methadone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Oral Methadone
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
The study was halted prematurely as it was very difficult to recruit participants. Of the 4 consented participants, none provided the information needed for any of the outcome measures, so no results are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT04941443/Prot_SAP_000.pdf